CLINICAL TRIAL: NCT04678635
Title: Chronic Transcranial Direct Current Stimulation in Patients With Systemic Autoimmune Myopathies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Samuel Katsuyuki Shinjo, PhD, Professor, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MYO-HCFMUSP-08
Record Dates: First submitted 2020-12-12; First posted 2020-12-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Myopathy
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo-controlled study with application or not of chronic transcranial direct current stimulation sessions - associated with aerobic exercises - in patients with systemic autoimmune myopathies.
Who Masked: Participant, Investigator
Masking Description: Double-blind study to transcranial direct current stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial direct current stimulation (Experimental): Transcranial direct current stimulation session: the energy of the anode (transcranial current stimulation) will have as its source a battery-powered DC generator and will be exerted by two electrodes measuring 5x7cm and attached to the head. The electrodes will be located of the primary motor cortex. The electrode with cathode will be positioned at contralateral to the dominant limb and the anode charged electrode will be positioned in the supraorbital region ipsilateral to the dominant limb. The active current of direct transcranial stimulation will be applied with the intensity of electric current of 2mA and density of 0.057 mA/cm2 with duration of 20 minutes. The stimulation will happen simultaneously to aerobic exercises for 20 minutes. Total number of stimulation associated with aerobic exercise sessions: 10
  Interventions: Other: Chronic transcranial direct current stimulation
- Placebo (Placebo Comparator): This group will not receive a transcranial direct current stimulation session. However, the patients will do aerobic exercises for 20 minutes. Total number of sham-stimulation associated with aerobic exercise sessions: 10
  Interventions: Other: Chronic transcranial direct current stimulation

INTERVENTIONS:
Other: Chronic transcranial direct current stimulation — Chronic transcranial direct current stimulation

SUMMARY:
Systemic autoimmune myopathies are rheumatic diseases that affect the striatum skeletal muscles. The transcranial direct current stimulation technique has been frequent, for example, in patients with ischemic stroke or for the optimization of muscular performance in athletes. However, to date, there are no studies evaluating this technique in patients with systemic autoimmune myopathies. Therefore, the main objective of the present prospective, randomized, double-blind, placebo-controlled study is to evaluate the safety and efficacy of the application of chronic transcranial direct current stimulation sessions - associated with aerobic exercises - in the patients with systemic autoimmune myopathies.

DETAILED DESCRIPTION:
Systemic autoimmune myopathies are rheumatic diseases that affect the striatum skeletal muscles. Depending on the clinical, pathophysiological and laboratory characteristics, they may be subdivided into polymyositis, dermatomyositis, antissintetase syndrome, immune-mediated necrotizing myopathy, and among others. Recently, the literature has been presenting better pharmacological treatment options to control these diseases. Despite these advances, this group of diseases still continues to be associated with high morbidity and functional disability, mainly due to the proximal muscular weakness of the scapular and pelvic girdles that may prevent the total recovery of these patients. On the other hand, the association of the transcranial current stimulation technique with motor recovery has been frequent, for example, in patients with ischemic stroke or for the optimization of muscular performance in athletes. However, to date, there are no studies evaluating this technique in patients with systemic autoimmune myopathies. Therefore, the main objective of the present prospective, randomized, double-blind, placebo-controlled study is to evaluate the safety and efficacy of the application of chronic transcranial current stimulation session - associated with aerobic exercises - in patients with systemic autoimmune myopathies.

ELIGIBILITY:
Inclusion Criteria:

* Classification criteria - EULAR/ACR 2017
* Classification critera - Connors et al.

Exclusion Criteria:

* Neoplasia
* Using heart pacemarker
* Using visceral metalic clips
* Infections (HIV, HTLV-1, Hepatitis, etc)
* Pregnance
* Previous historical of convulsions or epilepsies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes Participant eligibility is based on self-representation of gender identity
Enrollment: 40 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-emergent advser events | After 30 minutes of intervention
  Frequency of disease relapses (based on the questionnaire of secondary outcome measures) and tolerability (patients' symptom registration)
Frequency of treatment-emergent adverse events [safety and tolerability] | Before stimulation
  Frequency of disease relapsing (based on the questionnaire of secondary outcome measures) and tolerability (patients' symptom registration)
Frequency of treatment-emergent adverse events [safety and tolerability] | Immediately after all stimulation section
  Frequency of disease relapsing (based on the questionnaire of secondary outcome
Frequency of treatment-emergent adverse events [safety and tolerability] | After 30 days after last stimulation section
  Frequency of disease relapsing (based on the questionnaire of secondary outcome
Frequency of treatment-emergent adverse events [safety and tolerability] | After 60 days after last stimulation section
  Frequency of disease relapsing (based on the questionnaire of secondary outcome
Frequency of treatment-emergent adverse events [safety and tolerability] | After 90 days after last stimulation section
  Frequency of disease relapsing (based on the questionnaire of secondary outcome
Frequency of treatment-emergent adverse events [safety and tolerability] | After 300 days after last stimulation section
  Frequency of disease relapsing (based on the questionnaire of secondary outcome

SECONDARY OUTCOMES:
Myositis Disease Activity Assessment Visual Analogue Scales (MYOACT) | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  This partially validated tool measures the degree of disease activity of extra-muscular organ systems and muscle. The questionnaire is a series of physician's assessments of disease activity. Score ranges: 0 (best) - 60 (worst).
Serum levels of Muscle enzymes | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  This partially validated tool measures the serum activities of at least 2 of the 4 muscle-associated enzymes including creatine phosphokinase (CK), the transaminases (ALT, AST), lactate dehydrogenase (LD) and aldolase. The reference range value of each muscle enzyme will depend on the laboratory anaysis (kits). International Unit: U/L.
Health Assessment Questionnaire (HAQ) | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  Especific questionnaire (health assessment questionnaire). Pontuaction 0.00 (best) - 3.00 (worst)
Manual Muscle Testing (MMT) | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  This partially validated tool assesses muscle strength using manual muscle testing (MMT). A 0 - 10 point scale is proposed for use. An abbreviated group of 8 proximal, distal, and axial muscles performs similarly to a total of 24 muscle groups, and is also proposed for use for research studies. Pontuaction: 0 (worst) - 80 (best)
Patient Global Activity | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  This partially validated tool measures the global evaluation by the patient, or by the parent if the patient is a minor, of the patient's overall disease activity at the time of assessment using a 10 cm. visual analogue scale. Pontuaction: 0 (best) - 10 (worst)
Physician Global Activity | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  This partially validated tool measures the global evaluation by the treating physician of the overall disease activity of the patient at the time of assessment using a 10 cm. visual analogue scale. Pontuaction: 0 (best) - 10 (worst)
Fatigue Severity Scale | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  The questionnaire offers general fatigue scored by the patients, from 0 (better) to 10 (worse).
Short Form McGill Pain Questionnaire 2 (SF-MPQ-2) | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  The questionnaire offers general pain scored by the patients, from 0 (better) to 10 (worse).
Short Physical Performance Battery (SPPB) | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  The value ranges from 0 to 4 in different aspects of funcionality. The scores are compared among different periods of intervention (real or sham-stimulation)
Timed up and go test | Six times: (a) Before stimulation; (b) Immediately after all stimulation section; (c) after 30, 60, 90 and 300 days after last stimulation section
  To determine fall risk and measure the progress of balance, sit to stand and walking (seconds). The duration will be compared to before versus after intervation (real or sham-stimulation). Long duration (worse) versus short duration (better)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel K Shinjo, Principal Investigator — Brazil
Locations (1):
- Samuel K Shinjo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Misse RG, Dos Santos AM, Borges IBP, Grecco MV, Faria MSMS, da Silva LRS, Correia BL, Kim AWS, Tanaka C, Greve JMD, Baptista AF, Shinjo SK. Impact of Transcranial Direct Current Stimulation in Pain, Fatigue, and Health Quality of Life of Patients with Idiopathic Inflammatory Myopathies: A Randomized, Double-Blind, Sham-Controlled Crossover Clinical Trial. Int J Rheumatol. 2024 Feb 1;2024:1583506. doi: 10.1155/2024/1583506. eCollection 2024. PMID 38332984